CLINICAL TRIAL: NCT05194176
Title: The Effect of Virtual Reality on Pulmonary Recovery and Mobility in Patients With Blunt Chest Trauma
Acronym: VIREX PURE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion rate too low.
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112814
Record Dates: First submitted 2022-01-02; First posted 2022-01-18 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Blunt Chest Trauma
Keywords: Virtual Reality; Trauma; Pulmonary Recovery
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will receive usual care. Patients will be instructed to perform respiratory exercises 8 times daily for 10 minutes and to extend these exercises 2 times daily with (sitting) physical exercises for an additional 10 minutes. Respiratory exercises include using incentive spirometry and exercises for deep breathing, huffing and coughing. Patients receive a leaflet with the exercises described and the exercises will be performed once daily under supervision of a physiotherapist. The other sessions will be unsupervised.
- Virtual Reality (Experimental): The intervention group will be instructed to perform the respiratory exercises using the VR-intervention 8 times daily for 10 minutes and to extend these exercises 2 times daily with (sitting) physical exercises for an additional 10 minutes. The respiratory exercises in VR are comparable to the exercises in usual care but performed in a virtual environment and without incentive spirometry. The physical exercises consist of several games through which patients are challenged to reach out to objects while engaging their core. Patients are allowed to continue these exercises or play some relaxation games for up to 30 minutes per session in total. The exercises will be performed once daily under supervision of a physiotherapist. The other sessions will be unsupervised.
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — For all VR exercises a head mounted display (HMD), the PICO G2 4K (Barcelona, Spain) will be used. Together with SyncVRMedical (Utrecht, Netherlands) a VR dashboard has been created from which patients can chose the different exercises.
  Arms: Virtual Reality

SUMMARY:
Blunt chest trauma comprises over 10% of all trauma patients presenting to emergency departments worldwide and is the most frequent injury in polytrauma patients. It is associated with high risk (>10%) of pulmonary complications such as pneumonia. Pillars of treatment are adequate pain relief, respiratory function exercises and rapid mobilisation through physiotherapy. Inadequate pain control can result in restricted ventilatory function and in reduced mobility, both resulting in a higher risk of particularly pulmonary complications. Virtual Reality (VR) might be an easy to use, individualized, and harmless technique that can facilitate pulmonary recovery and aid in the prevention of complications through reducing pain and promoting exercising. The investigators hypothesize that VR improves respiratory function and mobilisation in the post-acute phase of blunt chest trauma by distracting patients from pain and stress, and by stimulating pulmonary and physical exercise.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the trauma ward with sustained blunt chest trauma
* Age≥16
* Patient is willing and able to comply with the study protocol

Exclusion Criteria:

* Neurotrauma with GCS ≤13
* History of dementia, seizures, epilepsy
* Severe hearing/visual impairment not corrected
* Head wounds or damaged skin with which comfortable and hygienic use is not possible.
* Stay at intensive care unit (ICU) during current hospital admission.
* Erect position in bed not possible/allowed.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Inspiration volume, mean change from baseline | From baseline to end of treatment at day 5.
  Mean change from baseline in inspiration volume in ml, measured with an incentive spirometer (Voldyne)
Inspiration volume, repeated measures over 5 days | Twice daily from enrollment to day 5 of treatment
  change in mean daily inspiration volume in mL, measured with an incentive spirometer (Voldyne)

SECONDARY OUTCOMES:
Time spent sitting or standing, mean change from baseline | Continuously from enrollment to end of treatment at day 5.
  Measured continuously using a wearable activity monitor, calculated as percentage of time spent sitting or standing.
Length of hospital stay | At end of follow-up, 30 days after discharge
  Length of hospital stay in days
Pulmonary complications during admission | At end of follow-up, 30 days after discharge
  Number and type of pulmonary complications during admission
Transfers to ICU | At end of follow-up, 30 days after discharge
  Participant transferred to ICU during admission yes/no?
Readmission within 30 days | At end of follow-up, 30 days after discharge
  Participant readmitted within 30 days, yes/no
Pain score during breathing exercise using Visual Analogue Score (VAS) | Daily from baseline to end of treatment at day 5.
  VAS pain score during breathing exercise (0-100mm). A higher score means a worse outcome.
Powerless in Daily living questionnaire | Daily from baseline to end of treatment at day 5.
  Powerless in Daily living questionnaire (0-21), a higher score means a worse outcome.
Quality of Recovery-15 questionnaire | Daily from baseline to end of treatment at day 5.
  Quality of Recovery-15 questionnaire (0-150), a higher score means a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable patient characteristics, questionnaire data, diaries and measurements will be shared in a pseudonimised manner in DANS EASY under restricted access
Supporting Information: SAP, Analytic Code

REFERENCES:
- [Derived] Groenveld TD, Smits IG, Scholten N, de Vries M, van Goor H, Stirler VM. Pulmonary and Physical Virtual Reality Exercises for Patients With Blunt Chest Trauma: Randomized Clinical Trial. JMIR Serious Games. 2024 Dec 9;12:e54389. doi: 10.2196/54389. PMID 39652866